CLINICAL TRIAL: NCT05653258
Title: Single Nuclei RNA-sequencing to Map Adipose Cellular Populations and Senescent Cells in Older Subjects
Brief Title: Single Nuclei RNA-seq to Map Adipose Cellular Populations and Senescent Cells in Older Subjects
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Nicolas Musi, MD, Staff Physician IV, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00002506; R01AG075684 (NIH)
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Healthy Lifestyle
Keywords: Lifestyle intervention; Single RNA sequencing; Cell Senescence
MeSH Terms: conditions — Obesity | interventions — Exercise; Diet; Dasatinib; Quercetin

STUDY DESIGN:
Intervention Model Description: All participants will undergo cellular/molecular profiling and older obese participants will be randomized into 3 arms.
Who Masked: Participant, Investigator
Masking Description: Investigators and subjects randomized to study drug/placebo will be blinded to which intervention they receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Younger Lean Group (Other): Participants will be aged 18-30 years and have a BMI of 18.5 - 24.9 kg/m2
  Interventions: Procedure: Abdominal adipose tissue biopsy
- Older Lean Group (Other): Participants will be over 65 years of age with a BMI of 18.5 to 24.9 kg/m2
  Interventions: Procedure: Abdominal adipose tissue biopsy
- Older Obese Group (Experimental): Participants will be over 65 years of age with a BMI of 30-39.9 kg/m2.
  Interventions: Other: Lifestyle Intervention; Drug: Dasatinib 100 MG; Drug: Quercetin 1000mg; Drug: Placebo; Procedure: Abdominal adipose tissue biopsy
- Younger Obese Group (Experimental): Participants will be ages 18-30 years and have a BMI OF 30.0-39.9 kg/m2
  Interventions: Procedure: Abdominal adipose tissue biopsy

INTERVENTIONS:
Other: Lifestyle Intervention — 1. Exercise: Subjects will undergo a combined aerobic and resistance exercise intervention. The investigators propose a multi-modal training program because they improve metabolic outcomes and adding resistance training reduces the risk of muscle loss during weight loss. Subjects will exercise in the gym for three sessions per week for 10 weeks under supervision of an exercise physiologist. On each session, aerobic exercise will be followed by resistance exercise.
  2. Diet: The aim of the dietary intervention is to reduce caloric intake sufficient to result in 8-10% weight loss, while incorporating behavioral and dietary strategies to maximize adherence and to minimize risk of muscle and bone loss. Subjects will attend small-group sessions led by a dietitian for changing their dietary composition to follow American Heart Association (AHA)/American College of Cardiology (ACC) guidelines.
  Other Names: Exercise and Diet
  Arms: Older Obese Group
Drug: Dasatinib 100 MG — 100 mg of dasatinib (D) daily for 3 consecutive days plus quercetin (Q) for the same 3 consecutive days, followed by a 25-day (+/- 2 day) no-drug period to complete a single round. This will be repeated twice more until completing 3 rounds total in approximately 10 consecutive weeks.
  Other Names: Sprycell
  Arms: Older Obese Group
Drug: Quercetin 1000mg — Quercetin (Q) (4) 250 mg capsules daily (total 1000 mg daily) plus dasatinib (D) same 3 consecutive days, followed by a 25-day (+/- 2 day) no-drug period to complete a single round. This will be repeated twice more until completing 3 rounds total in approximately 10 consecutive weeks.
  Arms: Older Obese Group
Drug: Placebo — Subjects will receive a placebo (methylcellulose) to provide a similar mass, number of tablets/ capsules, and frequency as the senolytic arm.
  Other Names: Placebo capsule
  Arms: Older Obese Group
Procedure: Abdominal adipose tissue biopsy — All participants will undergo baseline biopsies of subcutaneous abdominal adipose tissue for cellular/molecular profiling via snRNA-seq
  Other Names: Subcutaneous abdominal adipose tissue biopsy

SUMMARY:
All participants will undergo baseline biopsies of subcutaneous abdominal adipose tissue for cellular/molecular profiling via snRNA-seq and metabolic/physiological assessments (insulin sensitivity, glucose tolerance, and β-cell function). Older obese participants will be randomized into three arms: lifestyle intervention (n=24), senolytics (n=24), or placebo (n=24).

DETAILED DESCRIPTION:
All participants after consent and enrollment will undergo adipose tissue single nuclei RNA sequencing and metabolic phenotyping. Subjects will undergo glucose tolerance testing to document glucose tolerance status. Each subject will be provided an accelerometer to be worn on their dominant wrist for 7 days for assessment of habitual activity.

A dietitian will teach them to utilize the SmartIntake3 smartphone food picture application (app) for a 7-day food record. The app will be used to record amount of each meal consumed in order to determine daily food and beverage and supplement intake and quantity for dietary composition analysis. DEXA analysis will be performed to measure lean and fat body mass.

Subjects will undergo evaluation of physical function/performance, including the Short Physical Performance Battery (SPPB) and VO2 peak testing for assessment of aerobic capacity. The SPPB will be done in older adults only.

The NIH Patient-Reported Outcomes Measurement System (PROMIS) will be used to measure participants' self-report of symptoms, function, and health-related quality of life in the domains of physical, mental and social health.

All subjects will undergo a two-step euglycemic insulin clamp and indirect calorimetry.

Only older obese participants will continue to the randomization to likestyle intervention, senolytic agents or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Both Sexes
2. Age: younger lean group 18-30 years with BMI 18.5-24.9 kg/m2; younger obese group 18-30 with BMI 30.0 -39.9; older obese group ≥ 65 years with BMI 30.0-39.9
3. All races and ethnic groups
4. Community dwelling
5. Sedentary (≤1.5 h of exercise per week)
6. Nondiabetic (fasting plasma glucose < 126 mg/dl, 2-h glucose during oral glucose tolerance test (OGTT) < 140mg/dl, and A1c < 6.5%
7. For all female participants who are women of childbearing potential (WOCBP), who are not pregnant or breast feeding, at least one of the following conditions must apply:

   A documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy Use of a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency (implantable progesterone-only hormone contraception, intrauterine hormone releasing system, bilateral tubal occlusion, vasectomized partner) during the intervention period of the study and for at least 30 days after the last dose of study intervention to eliminate any reproductive safety risk of the study drug.

   Use of a contraceptive method that is highly effective (with a failure rate of <1% per year), with high user dependency, (oral/intravaginal/injectable combined estrogen and progesterone contraception, oral/injectable progesterone only hormone contraception, sexual abstinence) during the intervention period and for at least 30 days after the last dose of study intervention to eliminate any reproductive safety risk of the study drug. In addition to the highly effective methods: male or female condom with or without spermicide; cervical cap, diaphragm, or sponge with spermicide; a combination of male condom with either cervical cap, diaphragm, or sponge with spermicide.
8. ECG value after 10 minutes of resting in the supine position in the following ranges:

120ms<PR<220ms: QRS<120ms; QTc<430ms for males and QTc<450ms for females and normal ECG tracing, unless the investigator considers the ECG abnormality to be not clinically relevant.

Exclusion Criteria:

1. Diabetes, clinically diagnosed or HbA1c > 6.5% and/or fasting plasma glucose > 126 mg/dl and/or use of anti-diabetic medications.
2. Participating in > 1.5 h of structured exercise/week
3. Unstable weight (>3% change in last 3 months)
4. Neurological, musculoskeletal, or other conditions that may limit subject's ability to complete study physical assessment and training
5. Active autoimmune/inflammatory disease including: rheumatoid arthritis, multiple sclerosis, systemic lupus erythematous, inflammatory bowel disease
6. Laboratory parameters outside the normal range:

   * impaired kidney function (eGFR < 30ml/min/1.73m² as calculated by the CKD-EPI equation);
   * impaired liver function (AST or ALT level > 2 times upper limit of normal (ULN);
   * total Bilirubin level > 1.5 times ULN;
   * TSH > 1.5 times ULN or < lower limit of normal (LLN);
   * Hemoglobin <10.0 g/dl; Platelets <125,000 cell/mm³;
   * Platelets < 125,000 cell/mm³
   * Prothrombin time (PT) > 1.0 times ULN
   * Partial prothrombin time (PTT) > 1.0 times ULN.
7. Active gastrointestinal disease; coagulopathy; GI bleed within 6 months
8. Clinically significant heart disease (e.g. NYH Classification >II; ischemia)
9. Peripheral vascular disease (claudication)
10. QTc prolongation >45 msec
11. Use of anti-arrhythmic medications known to cause QTc prolongation, anti-platelet or anti-coagulant medication (see section 5.3)
12. Use of quinolone antibiotics or any other drugs that may prolong the QTc interval (see section 5.3)
13. Pulmonary disease (COPD), severe asthma or exercise-induced asthma
14. Recent systemic or pulmonary embolus
15. Uncontrolled blood pressure (systolic BP>170, diastolic BP>95 mmHg)
16. Smoking, alcohol use (history of regular alcohol consumption exceeding 7 drinks/week for female participants or 14 drinks/week for male participants. 1 drink = 5 ounces [150ml] of wine or 12 ounces [360ml] of beer or 1.5 ounces [45ml] of hard liquor) or recreational drug use (other than marijuana)
17. Pregnant or breastfeeding
18. Postmenopausal women new (within 6 months) to systemic hormone replacement therapy
19. Previous bariatric surgery
20. History of stroke with motor disability
21. Recent (3 years) treated cancer other than basal cell carcinoma
22. Acute or chronic infection
23. Medication that might interfere with metabolic studies (weight loss medication, systemic steroids, immunosuppressants) within 6 months (see section 5.3)
24. Potentially senolytic agents within the last 6 months: fisetin, quercetin, luteolin, dasatinib, piperlongumine, or navitoclax (see section 5.3)
25. History of allergy to dasatinib, quercetin and/or lidocaine.
26. Concurrent enrollment in another interventional trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | Week 4 and Week 15
  Change in skeletal muscle insulin sensitivity
Glucose tolerance | Baseline to Week 14
  Measurement of change in glucose tolerance using a glucose tolerance test

SECONDARY OUTCOMES:
Senescence-associated secretory phenotype (SASP) | Baseline to Week 16
  Measurement of change of SASP in adipose tissue

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Musi, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Unidentified data will be shared Research findings will be published in peer-reviewed scientific journals and will be presented at scientific meetings. Data derived from this study will be available upon request to regulatory bodies including NIH, UTHSCSA, DSMB, and the IRB.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available after study completion and analysis.